CLINICAL TRIAL: NCT03823625
Title: SQUINT (Squamous Immunotherapy Nivolumab-Ipilimumab Trial): An Open-label, Randomized, Parallel, Non Comparative, Phase II Trial of Nivolumab Plus Ipilimumab Versus Platinum-based Chemotherapy Plus Nivolumab in Chemonaive Metastatic or Recurrent Squamous-Cell Lung Cancer (SqLC)
Brief Title: An Open-label, Randomized, Parallel, Non Comparative, Phase II Trial of Nivolumab Plus Ipilimumab Versus Platinum-based Chemotherapy Plus Nivolumab in Chemonaive Metastatic or Recurrent Squamous-Cell Lung Cancer (SqLC)
Acronym: SQUINT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Ricerca Traslazionale (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SQUINT-FoRT 04
Record Dates: First submitted 2018-02-02; First posted 2019-01-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Squamous-Cell Lung Cancer
Keywords: SqLC
MeSH Terms: interventions — Nivolumab; Ipilimumab; Platinum Compounds

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARM A: Nivolumab plus Ipilimumab (Experimental): Immunotherapy will be given up to disease progression, toxicity or patient refusal and in any case for up to 24 months. Platinum-based chemotherapy will be given up to 6 cycles.
  Interventions: Drug: Nivolumab plus Ipilimumab
- ARM B: Platinum-based chemotherapy plus Nivolumab (Experimental): Platinum-based chemotherapy will be given up to 6 cycles. Immunotherapy will be given up to disease progression, toxicity or patient refusal and in any case for up to 24 months.
  Interventions: Drug: Platinum-based chemotherapy plus Nivolumab

INTERVENTIONS:
Drug: Nivolumab plus Ipilimumab — Nivolumab will be administered at the standard dose of 360 mg every 3 weeks. Ipilimumab will be administered at the dose of 1 mg/kg every 6 weeks.
  Arms: ARM A: Nivolumab plus Ipilimumab
Drug: Platinum-based chemotherapy plus Nivolumab — Nivolumab will be administered at the standard dose of 360 mg every 3 weeks.
  Platinum-based chemotherapy will be chosen by the investigator among the following regimens:
  * Cisplatin 80 mg/mq iv day 1 and Gemcitabine 1250 mg/mq iv days 1 and 8 every 21 days;
  * Carboplatin AUC 5 iv day 1 and Gemcitabine 1000 mg/mq iv days 1 and 8 iv every 21 days;
  * Carboplatin AUC 6 iv day 1 and paclitaxel 200 mg/mq iv day 1 every 21 days.
  Arms: ARM B: Platinum-based chemotherapy plus Nivolumab

SUMMARY:
Non-small-cell Lung Cancer (NSCLC) remains the leading cause of cancer death in Western Countries. Approximately 85% of lung cancers are of the non-small-cell type (NSCLC), with 25-30% of NSCLC being squamous histology type. Unlike nonsquamous NSCLC, squamous NSCLC rarely harbors epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) mutations for which there are directed therapies, and until the recent approval of immunotherapies for pretreated squamous NSCLC, a limited number of traditional cytotoxic chemotherapy drugs have been FDA-approved for use in the treatment of advanced and metastatic squamous NSCLC. A platinum-based combination chemotherapy regimen has been the standard first-line treatment for all NSCLC. Carboplatin is frequently substituted for cisplatin for patients who have poor renal function or who experience toxicities from cisplatin (most notably, nausea and vomiting). Taxanes, especially paclitaxel, or vinorelbine or gemcitabine, commonly complete the standard two-drug backbone of platinum-based chemotherapy for the first-line treatment of NSCLC, with platin-gemcitabine as the most commonly used regimen in Europe in patients with squamous-histology. A recent press release announced that pembrolizumab plus chemotherapy produced higher response rate when compared to chemotherapy alone in patients with squamous-cell lung cancer. Nevertheless, no data on Progression-Free Survival (PFS) and Overall Survival (OS) are available. Therefore, considering the lack of data in patients with squamous histology and the lack of information about efficacy of combinations of immune-checkpoints inhibitors versus immune-checkpoint inhibitor plus chemotherapy, there is a strong rationale for conducting a study assessing efficacy of such strategies in patients with advanced, metastatic squamous-cell lung cancer.

DETAILED DESCRIPTION:
Better understanding of the role of the immunological system in tumor control has opened multiple doors to implement different strategies to enhance immune response against cancer cells. It is known that tumor cells elude immune response by several mechanisms. The development of monoclonal antibodies against the checkpoint inhibitor programmed cell death protein 1 (PD-1) and its ligand (PD-L1), on T cells, has led to high activity in cancer patients with long lasting responses. In the KEYNOTE 024 the anti-PD-1 inhibitor Pembrolizumab significantly prolonged progression-free survival (PFS) and overall survival (OS) of patients with advanced NSCLC and high PD-L1 level (>50% of tumor cells) compared to platinum based chemotherapy, thus becoming a new standard of care in front line setting. However, the trial was not restricted to squamous population, with approximately 18% per arm having this histology. Nivolumab, another PD-1 inhibitor, has been recently approved for the treatment of squamous cell lung cancer patients, given the survival advantage demonstrated in a phase III trial comparing the drug to docetaxel, in second-line setting. Importantly, the benefit produced by the drug was irrespective of PD-L1 expression suggesting that the high mutation burden of squamous-cell lung carcinoma is more relevant than the expression of a single biomarker, at least in pretreated individuals. In addition, recent studies in chemo naive patients with non-squamous histology demonstrated that combination of chemotherapy and immunotherapy is superior to chemotherapy alone in terms of Overall Survival irrespective of PD-L1 expression (Keynote 189 and IMPOWER 150). In addition, the CheckMate 227 study recently showed that, in chemonaive NSCLC, combination of nivolumab and ipilimumab was superior to chemotherapy alone in patients with high tumor mutational burden (TMB), irrespective of PD-L1 expression. A recent press release announced that pembrolizumab plus chemotherapy produced higher response rate when compared to chemotherapy alone in patients with squamous-cell lung cancer (Keynote 407). Nevertheless, no data on Progression-Free Survival and Overall Survival are available. Therefore, considering the lack of data in patients with squamous histology and the lack of information about efficacy of combinations of immune-checkpoints inhibitors versus immune-checkpoint inhibitor plus chemotherapy, there is a strong rationale for conducting a study assessing efficacy of such strategies in patients with advanced, metastatic squamous-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients willing and able to give written informed consent;
* Histologically confirmed diagnosis of Stage IIIB-not amenable to radical treatment or Stage IV or recurrent squamous-cell lung carcinoma;
* Tumor p63 (or p40) positive and TTF1 negative;
* Availability of tumor tissue for PD-L1 expression analysis. One formalin-fixed paraffin embedded tumor tissue block or a minimum of 16 unstained tumor tissue sections are acceptable. The tumor tissue sample may be fresh or archival if obtained within 6 months prior to enrollment, and there can have been no systemic therapy (eg, adjuvant or neoadjuvant chemotherapy) given after the sample was obtained. Tissue must be a core needle biopsy, excisional or incisional biopsy. Fine needle biopsies or drainage of pleural effusions with cytospins are not considered adequate for biomarker review. Biopsies of bone lesions that do not have a soft tissue component or decalcified bone tumor samples are also not acceptable;
* Availability of PD-L1 status;
* Chemonaive patient. Adjuvant/neoadjuvant chemotherapy is allowed if therapy was completed at least 6 months before trial inclusion;
* Performance status 0-1 (ECOG);
* Patient compliance to trial procedures;
* Age ≥ 18 years;
* Written informed consent;
* Adequate BM function (ANC ≥ 1.5x109/L, Platelets ≥ 100x109/L, HgB > 9g/dl);
* Adequate liver function (bilirubin < G2, transaminases no more than 3xULN/<5xULN in present of liver metastases);
* Normal level of alkaline phosphatase and creatinine;
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of approved contraceptive method [intrauterine contraceptive device (IUD), birth control pills, or barrier device] during and for twenty-three (23) weeks after end of treatment;
* If men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product;
* Prior palliative radiotherapy to non-CNS lesions must have been completed at least 2 weeks prior to treatment. Patients with symptomatic tumor lesions that may require palliative radiotherapy within 4 weeks of first treatment are strongly encouraged to receive palliative radiotherapy prior to treatment. Patients are eligible if CNS metastases are adequately treated and patients are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to randomization;
* Patients must be either off corticosteroids, or on a stable or decreasing dose of ≥10 mg daily prednisone (or equivalent) for at least 2 weeks prior to randomization.

Exclusion Criteria:

* No tumor tissue available;
* Tumor negative for p63 (or p40) or positive for TTF1;
* Previous chemotherapy for stage IV disease;
* Adjuvant or neoadjuvant chemotherapy completed less than 6 months before trial inclusion; adjuvant or neoadjuvant immunotherapy is not allowed;
* Concomitant radiotherapy or chemotherapy;
* Untreated brain metastases;
* Diagnosis of any other malignancy during the last 2 years, except for in situ carcinoma of cervix uteri and cutaneous squamous cell carcinoma;
* Pregnancy or lactating;
* Other serious illness or medical condition potentially interfering with the study.

Nivolumab and ipilimumab specific exclusion

* Patients with an active, known or suspected autoimmune disease. Patients with type I diabetes mellitus; hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll;
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease;
* Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection;
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of Overall Survival in subjects with Stage IIIB not amenable to radical treatment or Stage IV or recurrent squamous-cell lung carcinoma treated in the study | 12 months
  Overall Survival rate at 12 months in Arm A and B

SECONDARY OUTCOMES:
Biomarkers analysis | 48 months
  Correlation of PD-L1 expression and/or TMB with outcome in Arm A and B
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 48 months
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cappuzzo, Principal Investigator — Ospedale di Ravenna
Locations (18):
- Italy (18):
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)- Oncologia Medica, Meldola, Forlì- Cesena
  - Ospedale "Infermi" Rimini, Rimini, Italia
  - Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture, Potenza
  - Sacro Cuore- Don Calabria Hospital- U.O.C. Oncologia Medica, Negrar, Verona
  - Istituto Toscano Tumori Ospedale San Donato- U.O.C. di Oncologia Medica Dipartimento di Oncologia USL-8, Arezzo
  - IRCCS A.O.U. San Martino- IST- Istituto Nazionale per la Ricerca sul Cancro- U.O.S. Tumori Polmonari, Genova
  - Istituto Europeo di Oncologia - Divisione di Oncologia Toracica, Milan
  - A.O.U. Policlinico di Modena- Oncologia Ematologia e Malattie Apparato Respiratorio, Modena
  - A.O.R.N dei Colli - Ospedale Monaldi, Napoli
  - I.R.C.C.S. Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo
  - Casa di Cura La Maddalena- U.O. Oncologia medica, Palermo
  - Azienda Ospedaliera di Perugia- S.C. Oncologia Medica, Perugia
  - Ospedale di Ravenna- Oncologia Medica, Ravenna
  - IRCCS Arcispedale Santa Maria Nuova, Reggio Emilia
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Policlinico Universitario "Campus Biomedico" di Roma, Roma
  - Policlinico 'G.B.Rossi' Borgo Roma - A.O.U. Integrata (Giampaolo Tortora)- Oncologia Medica, Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cappuzzo F, Ricciuti B, Delmonte A, Bonanno L, Wang X, Lye WK, Gortz A, Andrikou K, Dal Maso A, Minuti G, Papi M, Alessi JV, Di Federico A, Rodig S, Awad MM, Metro G, Attili I, Vitiello F, Pilotto S, Gori S, Rossi G, Buglioni S, Giannarelli D, Landi L. MAPK Pathway-Activating Alteration and Immunotherapy Efficacy in Squamous Cell Lung Carcinoma: Results from the Randomized, Prospective SQUINT Trial. Clin Cancer Res. 2025 Mar 17;31(6):1027-1036. doi: 10.1158/1078-0432.CCR-24-2077. PMID 39836372